CLINICAL TRIAL: NCT04433494
Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of TY-302 Capsules in Patients With Advanced Solid Tumors in China
Brief Title: A Study of TY-302 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYKM1602101
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer; Solid Tumor
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TY-302 ; TY-302 combine with Tamoxifen (Experimental): 1. TY-302
     * Find the maximum tolerated dose(MTD) and the recommended phase 2 dose (RP2D) of TY-302, given orally.
     * Increased dose cohorts from low dose to MTD, starting at 25mg daily.
  2. TY-302 combine withTamoxifen in dose-escalation stage
     * TY-302: RP2D-1to RP2D daily for 28 days of each 28 day cycle.
     * Tamoxifen: 20mg twice daily for 28 days of each 28 day cycle.
  3. TY-302 combine withTamoxifen in dose-expansion stage
     * TY-302: RP2D daily for 28 days of each 28 day cycle.
     * Tamoxifen: 20mg twice daily for 28 days of each 28 day cycle.
  Interventions: Drug: TY-302: capsule, 25mg/50mg ; Tamoxifen: tablet,10mg

INTERVENTIONS:
Drug: TY-302: capsule, 25mg/50mg ; Tamoxifen: tablet,10mg — TY-302 is taken orally. Tamoxifen is taken orally.
  Other Names: TY-302; Tamoxifen Citrate

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of TY-302 single and the combination with Tamoxifen in dose-escalation and dose-expansion study.The drugs involved in this study are:

* TY-302
* Tamoxifen

DETAILED DESCRIPTION:
This is an open-label, single-arm, phase I trial. The purpose of this study is to :

* Test a safe and tolerable dose of TY-302 single and the combination with Tamoxifen
* Determine the response rate of the combination
* Further evaluate the safety and side effect profile for the combination of TY-302 and Tamoxifen.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70years old, male or female with solid tumors, female with breast cancer
2. Histological or cytological confirmation diagnosis of advanced solid tumors (except small cell lung cancer and eye cancer) in TY-302 alone study; and advanced breast cancer in the combination study.
3. Biopsy proven diagnosis of ER and/or PR positive, HER2 negative.
4. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
6. Life expectancy of at least 3 month.
7. Adequate organ function as defined by the following criteria:

   Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤2.5 x upper limit of normal (ULN), or AST and ALT ≤5 x ULN if liver function abnormalities are due to underlying malignancy; total serum bilirubin ≤1.5 x ULN; Absolute neutrophil count (ANC) ≥1.5×109/L; platelets(PLT)≥75×109/L ; Hemoglobin(Hb) ≥ 90g/L; Serum creatinine ≤1.5 x ULN; Left ejection fraction (LVEF)≥50%; QTc≤470 msec (based on the mean value of the triplicate ECGs).
8. Female subjects have a negative urine or serum pregnancy.
9. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.

Exclusion Criteria:

Subjects presenting with any of the following were not to be included in the study:

1. Previously treated by other CDK4/6 inhibitor.
2. Hypersensitivity to TY-302(or Tamoxifen in the combination study) or to any of its excipients.
3. Ocular fundus diseases in the combination study.
4. Uncontrolled intercurrent illness including active infection, human immunodeficiency virus infection, active hepatitis or other severe acute or chronic medical or psychiatric condition.
5. Current alcohol/drug abuse or dependence.
6. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE grade≥2, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure of NCI CTCAE grade≥2, cerebrovascular accident.
7. Presence of a condition that would interfere with enteric absorption of TY-302 and/or Tamoxifen.
8. Any cytotoxic chemotherapy, investigational agents or anticancer drugs for the treatment from a previous treatment regimen within 4 weeks of the first dose.
9. Spinal cord compression or brain metastases unless asymptomatic.
10. Major surgery within 8 weeks of first study treatment.
11. Current use or anticipated need for drugs that are known strong CYP3A4 inhibitors, strong CYP3A4 inducers, Narrow therapeutic index for CYP3A sensitive substrates, CYP2D6 inhibitors, CYP2D6 inducers.
12. Patients on chronic anticoagulation.
13. The subject inappropriate for entry into this study in the judgment of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only femal can be included in breast cancer on the combination study.
Enrollment: 60 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of TY-302 | 1 year
  To determine the MTD and RP2D of TY-302 in subjects with solid tumors
Dose Limiting Toxicity (DLT) of TY-302 | First 35 days of dosing
  Incidence of Dose Limiting Toxicity (DLT) of TY-302
Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of TY-302 combine with Tamoxifen | 1 year
  To determine the MTD and RP2D of TY-302 and Tamoxifen on the combination in subjects with breast cancer
Dose Limiting Toxicity (DLT) of TY-302 combine with Tamoxifen | First 28 days of dosing
  Incidence of Dose Limiting Toxicity (DLT) of TY-302 and Tamoxifen on the combination
Overall Response Rate (ORR) of TY-302 combine with Tamoxifen | 6 months
  To assess the effect of TY-302 combine with Tamoxifen on ORR( the proportion of patients with a best overall response of complete response (CR) or partial response (PR) assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) ) in the treatment of ER+/HER2- advanced breast cancer.
Disease Control Rate(DCR) of TY-302 combine with Tamoxifen | 9 months
  To assess the effect of TY-302 combine with Tamoxifen on DCR(the proportion of patients with CR, PR, or stable disease(SD) assessment in accordance to RECIST 1.1) in the treatment of ER+/HER2- advanced breast cancer.
Duration of Response (DOR) of TY-302 combine with Tamoxifen | 9 months
  To assess the effect of TY-302 combine with Tamoxifen on DOR( the time from first documented response (PR or CR) to the date of first documented disease progression or death due to any cause determined by Investigator assessment in accordance to RECIST 1.1) in the treatment of ER+/HER2- advanced breast cancer.
Progression-free Survival (PFS) of TY-302 combine with Tamoxifen | 12 months
  To assess the effect of TY-302 combine with Tamoxifen on PFS(time from date of first dose of study treatment to date of first documented disease progression or death due to any cause determined by Investigator assessment in accordance to RECIST 1.1) in the treatment of ER+/HER2- advanced breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical Colledge
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical Colledge, Beijing, Beijing Municipality, China